CLINICAL TRIAL: NCT04798547
Title: Outcomes of Short-length vs Standard-length Myotomy Using Per-Oral Endoscopic Myotomy (POEM) for Achalasia: A Randomized Controlled Pilot Study
Brief Title: Short Vs Standard Length Myotomy in Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, A. Aziz Aadam, Associate Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00212053
Record Dates: First submitted 2021-02-05; First posted 2021-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Length Myotomy (Placebo Comparator): Patients randomized to received 8 cm standard length myotomy in Per-Oral Endoscopic Myotomy (POEM) for achalasia
  Interventions: Procedure: Standard Length Myotomy
- Short Length Myotomy (Experimental): Patients randomized to received 4 cm standard length myotomy in Per-Oral Endoscopic Myotomy (POEM) for achalasia
  Interventions: Procedure: Short Myotomy

INTERVENTIONS:
Procedure: Short Myotomy — Evaluation of short length myotomy
  Arms: Short Length Myotomy
Procedure: Standard Length Myotomy — Standard Length Myotomy
  Arms: Standard Length Myotomy

SUMMARY:
The objective of this randomized controlled trial (non-inferiority study) is to evaluate the outcomes of 4 cm short myotomy compared to the 8 cm standard length myotomy in Per-Oral Endoscopic Myotomy (POEM) for patients with achalasia. We hypothesize that a shorter myotomy with POEM will have the same clinical efficacy as standard length myotomy based on patient-reported Eckardt score with shorter procedure times and reduced complications.

DETAILED DESCRIPTION:
BACKGROUND:

Achalasia is a disorder of esophageal dysmotility characterized by dysfunctional peristalsis and increased lower esophageal sphincter (LES) tone. Achalasia is further divided into three subtypes using high-resolution manometry (HRM) following the Chicago Classification. Type I, or classic achalasia, and Type II achalasia are both characterized by aperistalsis and increased LES tone and are thought to be a spectrum of the same disease process with Type II evolving into Type I.

Per-oral Endoscopic Myotomy (POEM) was first developed in 2008 as a treatment for achalasia. The technique involves a trans-oral approach with a flexible endoscope. An endoscopic incision is made in the esophagus and a submucosal tract is created towards the LES and gastric cardia to expose the underlying muscle of the LES and distal esophagus. The inner circular muscle is then dissected to create a myotomy and the tract is then closed with endoscopic clips. By creating a myotomy, the increased LES tone is improved, allowing food to pass into the stomach in order to relieve the dysphagia caused by achalasia.

Unlike Type III achalasia, where POEM myotomy length is determined by HRM, the standard myotomy length in Type I/Type II achalasia is typically 8 cm. The rationale for the 8 cm myotomy is derived from the Heller myotomy procedure which is a laparoscopic surgery approach in which the teaching has been to perform at least a 5 cm myotomy in the esophagus and an additional 2-3 cm myotomy in the gastric cardia. However, the purpose of the myotomy in POEM, is to reduce the LES tone. The clinical efficacy of the procedure comes from the myotomy of the high pressure zone within the LES, which is only 2-3cm in length. This is much shorter than the current standard POEM myotomy length. There are a few potential pitfalls regarding longer myotomy lengths in the esophagus and in the gastric cardia. A longer esophageal myotomy may result in esophageal wall strain in the area weakened by esophageal myotomy resulting in a blown out myotomy which is identified by the presence of a pseudo-diverticulum endoscopically. Longer gastric cardia myotomy has been thought to lead to an increased rate of gastroesophageal reflux in patients undergoing POEM. There are no data looking at shorter myotomy lengths in POEM for Type I and Type II achalasia. Our anecdotal experience at Northwestern when performing short myotomy during POEM has not resulted in any difference in procedural efficacy.

STUDY ENDPOINTS:

Upon enrollment, patients will complete the Eckardt study questionnaire and the GERDQ questionnaire on the initial visit. Enrolled subjects will complete POEM as per clinical standard of care with the following specifications. Patients will be randomized to receive a short myotomy of 4 cm or standard myotomy of 8 cm. Following POEM, patients will be followed in clinic per standard of care and study questionnaires will be administered at follow-up visits. The Eckardt Symptom score is validated for research use in achalasia and is the tool with which we monitor success rates for treatment of achalasia. We will also monitor GERD symptoms with the GERDQ questionnaire. The endpoints for this study following randomization and completion of 30 POEM procedures are:

1. 3, 12 and 24-months of follow-up to monitor Eckardt score for all 30 participants
2. 3, 12 and 14-months of follow-up to monitor safety and GERD for all 30 participants

PROCEDURES INVOLVED:

Patients will be recruited from the pool of patients seen in esophageal clinics and endoscopy centers at Northwestern's Digestive Health Center who are specifically consented to undergo POEM for Type I or Type II achalasia and also in patients with EGJ outflow obstruction that demonstrate features of achalasia. Involvement with the study will not determine or affect eligibility or recommendation for POEM in the treatment of achalasia. Upon enrollment, patients will complete all study questionnaires on the initial visit - these include our GERDQ questionnaire and our Northwestern Esophageal Quality of Life Survey.

Following enrollment, 30 patients will be randomized to receive either a 4 cm or 8 cm myotomy. Randomization will occur via computer randomization software. At the time of the procedure, the endoscopist will be given the randomized grouping in an opaque envelope (either 4 cm or 8 cm myotomy). Participants will then undergo Per-Oral Endoscopic Myotomy as per standard of care with flexible endoscope using an anterior approach. The only difference in the procedure will be the length of the muscle layer dissection (myotomy). Fifteen subjects will undergo the standard 8 cm myotomy, which includes 7 cm myotomy of the esophagus and 1 cm myotomy of the gastric cardia. Fifteen subjects will undergo a short 4 cm myotomy, which includes 3 cm myotomy in the esophagus and a 1 cm myotomy of the gastric cardia. All participants will undergo intra-operative functional monitoring as is standard of care at Northwestern to ensure adequate response to myotomy. If the shorter myotomy is insufficient, the patient can undergo standard-length myotomy.

Participants will be monitored as per standard care before, during and after POEM procedure. Post-procedure follow-up for both groups will adhere to standard of care. Data will be collected on a prospective data from EPIC electronic health care records. Data collected will include demographic information, imaging results, functional studies (specifically EndoFlip and HRM) as well as questionnaire data.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18+ diagnosed with Type I or Type II achalasia, and patients with EGJ Outflow Obstruction with features of achalasia based on HRM or Endoscopic Functional Lumen Imaging Probe (EndoFLIP)
* All subjects must have given signed, informed consent prior to registration in the study

Exclusion Criteria:

* Patient with Type III achalasia or spastic esophageal dysmotility disorders requiring long myotomy as determined by HRM
* All patients who are unable or unwilling to give consent will not be included in the study
* Patients who are pregnant, vulnerable populations such as prisoners, life expectancy < 1 year based on concurrent comorbidities, coagulopathy with INR > 1.5 that cannot be reversed, thrombocytopenia with platelets < 50,000 that cannot be corrected with blood products, unable to safely undergo elective endoscopy due to current comorbidities, and inability to pass standard endoscope.
* Patients who have already undergone treatment with POEM or Heller Myotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Compare symptomatic improvement of achalasia based on Eckardt Score following POEM with 4 cm myotomy vs 8 cm myotomy | 2 years
  At 1, 6 and 12 months, patient reported outcome of achalasia symptoms will be assessed. The Eckardt Score is a validated research tool for achalasia symptoms. Scores range from 0-12. A higher score indicates worse symptoms. We will compare Eckardt Score pre-POEM and post-PEM at various time points.

SECONDARY OUTCOMES:
Compare procedure complications after 4 cm myotomy with POEM compared to 8 cm myotomy with POEM | 1 year
  We will monitor for any evidence of complications post-procedure including bleeding, perforation and blown-out myotomy.
Compare procedural time and intra-procedural findings between 4 cm myotomy with POEM compared to 8 cm myotomy with POEM | 1 year
  We will record procedure times and procedural findings including submucosal tunnel length, position of myotomy, cautery settings for myotomy, need for revision of myotomy and endoclips used for tunnel closure.
Compare post-POEM gastro-esophageal reflux between 4 cm myotomy and 8 cm myotomy using GERDQ assessment. | 2 years
  At 1, 6 and 12 months, patient reported outcome of acid reflux will be assessed. The GERDQ is a validated survey tool to assess acid reflux symptoms. Scores range from 0-18 with a higher score indicating worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen WF, Li QL, Zhou PH, Yao LQ, Xu MD, Zhang YQ, Zhong YS, Ma LL, Qin WZ, Hu JW, Cai MY, He MJ, Cui Z. Long-term outcomes of peroral endoscopic myotomy for achalasia in pediatric patients: a prospective, single-center study. Gastrointest Endosc. 2015 Jan;81(1):91-100. doi: 10.1016/j.gie.2014.06.035. Epub 2014 Aug 1. PMID 25088923
- [Result] Hungness ES, Sternbach JM, Teitelbaum EN, Kahrilas PJ, Pandolfino JE, Soper NJ. Per-oral Endoscopic Myotomy (POEM) After the Learning Curve: Durable Long-term Results With a Low Complication Rate. Ann Surg. 2016 Sep;264(3):508-17. doi: 10.1097/SLA.0000000000001870. PMID 27513156
- [Result] Laurino-Neto RM, Herbella F, Schlottmann F, Patti M. EVALUATION OF ESOPHAGEAL ACHALASIA: FROM SYMPTOMS TO THE CHICAGO CLASSIFICATION. Arq Bras Cir Dig. 2018;31(2):e1376. doi: 10.1590/0102-672020180001e1376. Epub 2018 Jul 2. PMID 29972404
- [Result] Taft TH, Carlson DA, Triggs J, Craft J, Starkey K, Yadlapati R, Gregory D, Pandolfino JE. Evaluating the reliability and construct validity of the Eckardt symptom score as a measure of achalasia severity. Neurogastroenterol Motil. 2018 Jun;30(6):e13287. doi: 10.1111/nmo.13287. Epub 2018 Jan 8. PMID 29315993
- [Result] Kahrilas PJ, Boeckxstaens G. The spectrum of achalasia: lessons from studies of pathophysiology and high-resolution manometry. Gastroenterology. 2013 Nov;145(5):954-65. doi: 10.1053/j.gastro.2013.08.038. Epub 2013 Aug 21. PMID 23973923
- [Result] Boeckxstaens GE, Zaninotto G, Richter JE. Achalasia. Lancet. 2014 Jan 4;383(9911):83-93. doi: 10.1016/S0140-6736(13)60651-0. Epub 2013 Jul 17. PMID 23871090
- [Result] Pandolfino JE, Kwiatek MA, Nealis T, Bulsiewicz W, Post J, Kahrilas PJ. Achalasia: a new clinically relevant classification by high-resolution manometry. Gastroenterology. 2008 Nov;135(5):1526-33. doi: 10.1053/j.gastro.2008.07.022. Epub 2008 Jul 22. PMID 18722376
- [Result] Spechler SJ, Castell DO. Classification of oesophageal motility abnormalities. Gut. 2001 Jul;49(1):145-51. doi: 10.1136/gut.49.1.145. PMID 11413123
- [Result] Pandolfino JE, Kahrilas PJ; American Gastroenterological Association. AGA technical review on the clinical use of esophageal manometry. Gastroenterology. 2005 Jan;128(1):209-24. doi: 10.1053/j.gastro.2004.11.008. No abstract available. PMID 15633138
- [Result] Kahrilas PJ, Katzka D, Richter JE. Clinical Practice Update: The Use of Per-Oral Endoscopic Myotomy in Achalasia: Expert Review and Best Practice Advice From the AGA Institute. Gastroenterology. 2017 Nov;153(5):1205-1211. doi: 10.1053/j.gastro.2017.10.001. Epub 2017 Oct 6. PMID 28989059
- [Result] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Result] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] Kane ED, Budhraja V, Desilets DJ, Romanelli JR. Myotomy length informed by high-resolution esophageal manometry (HREM) results in improved per-oral endoscopic myotomy (POEM) outcomes for type III achalasia. Surg Endosc. 2019 Mar;33(3):886-894. doi: 10.1007/s00464-018-6356-0. Epub 2018 Jul 27. PMID 30054739
- [Result] Li QL, Chen WF, Zhou PH, Yao LQ, Xu MD, Hu JW, Cai MY, Zhang YQ, Qin WZ, Ren Z. Peroral endoscopic myotomy for the treatment of achalasia: a clinical comparative study of endoscopic full-thickness and circular muscle myotomy. J Am Coll Surg. 2013 Sep;217(3):442-51. doi: 10.1016/j.jamcollsurg.2013.04.033. Epub 2013 Jul 25. PMID 23891074